CLINICAL TRIAL: NCT02197884
Title: An Open-Label, Fixed-Sequence Study to Assess Effects of Clarithromycin on the Single-Dose Pharmacokinetics of JNJ-54861911 in Healthy Male Subjects
Brief Title: A Study to Assess Effects of Clarithromycin on Pharmacokinetics of JNJ-54861911 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104763; 2014-001793-33 (EudraCT Number); 54861911ALZ1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54861911; Cytochrome P450 3A4 inhibitor; Itraconazole; Clarithromycin; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat; Itraconazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Itraconazole + JNJ-54861911 (Part 1) (Experimental): Single dose of JNJ-54861911, 25 milligram (mg) tablet orally on Day 1 and Day 9 along with itraconazole 200 mg (2*100 mg capsule) orally once daily from Day 5 to Day 12.
  Interventions: Drug: JNJ-54861911, 25 mg; Drug: Itraconazole 200 mg
- Clarithromycin + JNJ-54861911 (Part 2) (Experimental): Single dose of JNJ-54861911, 25 mg tablet orally on Day 1 and Day 9 along with clarithromycin 500 mg immediate release tablet orally twice daily from Day 5 to Day 12.
  Interventions: Drug: JNJ-54861911, 25 mg; Drug: Clarithromycin 500 mg

INTERVENTIONS:
Drug: JNJ-54861911, 25 mg — JNJ-54861911, 25 mg tablet orally on Day 1 and Day 9.
Drug: Itraconazole 200 mg — Itraconazole 200 mg (2*100 mg capsule) orally once daily from Day 5 to Day 12.
  Arms: Itraconazole + JNJ-54861911 (Part 1)
Drug: Clarithromycin 500 mg — Clarithromycin 500 mg immediate release tablet orally twice daily from Day 5 to Day 12.
  Arms: Clarithromycin + JNJ-54861911 (Part 2)

SUMMARY:
The purpose of this study is to assess the effects of strong cytochrome P450 (CYP) 3A4 inhibitors (Itraconazole and Clarithromycin), on pharmacokinetics (PK) (study of the way a drug enters and leaves the blood and tissues over time) of single dose of JNJ-54861911 in healthy male participants.

DETAILED DESCRIPTION:
This is a single-center, open-label (participants and researchers are aware about the treatment, participants are receiving), fixed-sequence study in healthy male participants consisting of 2 sequential parts. For all participants enrolled in either part, the study consists of 3 phases: Screening Phase (within 21 to 2 days prior to the first dose administration on Day 1), Open-label Treatment Phase (Day 1 up to Day 12), and Follow-up Phase (7 to 14 days after last dose administration). The maximum duration of study will be 7 weeks per participant. Study will be conducted in 2 parts to understand the relative role of CYP3A4 and amide hydrolysis pathways in JNJ-54861911 metabolism and any potential drug-drug interaction liability with inhibitors of these pathways. Itraconazole will be administered in Part 1 as mixed CYP3A4 and potential amide hydrolysis inhibitor. Clarithromycin will be administered in Part 2 as a pure CYP3A4 inhibitor. However, Part 2 of the study will only be conducted if a relevant interaction is observed with itraconazole based on an interim review of Part 1 data. Participants enrolled in Part 1 will receive single dose of JNJ-54861911, 25 milligram (mg) tablet orally on Day 1 and Day 9 along with itraconazole 200 mg (2*100 mg capsule) orally once daily from Day 5 to Day 12. Participants enrolled in Part 2 will receive single dose of JNJ-54861911, 25 mg tablet orally on Day 1 and Day 9 along with clarithromycin 500 mg immediate release tablet orally twice daily from Day 5 to Day 12. Blood samples will be collected pre-dose (Day 1) up to Day 13 to understand the PK characteristics of JNJ-54861911 and diaminothiazine (DIAT, a metabolite formed after amide hydrolysis of JNJ-54861911). In addition, a blood sample will be collected on Day -1 from all enrolled participants to study genotyping of CYP3A4 gene and other genetic factors that may influence the PK, safety, and/or tolerability of JNJ-54861911 and CYP3A4 inhibitors. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study, and are willing to participate in the study
* Body mass index between 18 and 30 kilogram per square meter
* Must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening or admission (up to Day 1 predose)
* Man, who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator, and must also agree to not donate sperm during the study and for 90 days after receiving the study drug
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening and/or admission and as per investigator's judgment

Exclusion Criteria:

* History of or current liver or renal impairment, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, dermatological or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to JNJ-54861911 or its excipients, itraconazole (Part 1 only) or clarithromycin (Part 2 only)
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening
* History of drug or alcohol abuse within 6 months before Screening or positive test result(s) for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines, benzodiazepines and cotinine) at Screening or admission
* Smoking of cigarettes (or equivalent) and/or used nicotine based products within 3 months prior to study drug administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-54861911 and diaminothiazine (DIAT) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Concentration (Tmax) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  The Tmax is time to reach the maximum observed plasma concentration.
Time to Last Quantifiable Plasma Concentration (Tlast) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  The Tlast is time to last observed quantifiable plasma concentration (Clast).
Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  The AUC (0-last) is area under the plasma concentration-time curve from time zero to time of last quantifiable concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Extrapolated Infinite Time (AUC [0-infinity]) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to extrapolated infinite time, calculated as the sum of AUC (0-last) and Clast/lambda(z), where AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time; Clast is the last observed quantifiable concentration; and lambda(z) is first-order rate constant associated with the terminal portion of the semilogarithmic drug concentration-time curve.
Area Under the Plasma Concentration-time Curve From Time Zero to Time 24 Hours (AUC [0-24]) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  Area under the plasma concentration-time curve from time zero to time 24 hours.
Elimination Half-Life (t1/2) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve, is calculated as 0.693 divided by lambda(z), where lambda(z) is first-order rate constant associated with the terminal portion of the curve. The t1/2 is the measure of time, for plasma concentration to decrease by one half.
Elimination Rate Constant (lambda[z]) of JNJ-54861911 and DIAT | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 18, 24, 36, 48, 72, 96 hours post-dose on Day 1 and 9
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the semilogarithmic drug concentration-time curve.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to follow-up (7 to 14 days after last dose administration)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; and congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium